CLINICAL TRIAL: NCT07383064
Title: Single Versus Multiple Vessels Endovascular Tibial Arteries Revascularization for Critical Limb Ischemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Mohammed Zakria Mohammed El Amir, Vascular surgery resident, Aswan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Asw.uni./980/9/24
Record Dates: First submitted 2026-01-16; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2024-12

CONDITIONS: Critical Limb Ischemia; Tibialis Vessels Occlusion
Keywords: Endovascular Revascularization for critical limb ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Single tibial artery Endovascular Revascularization (Active Comparator): Who undergo single tibial artery Endovascular Revascularization
  Interventions: Procedure: Endovascular Revascularization
- Multiple tibialis vessels Endovascular Revascularization (Sham Comparator): Who undergo more than one tibial artery Revascularization
  Interventions: Procedure: Endovascular Revascularization

INTERVENTIONS:
Procedure: Endovascular Revascularization — One would undergo single tibial artery Endovascular Revascularization
  Other Names: Endovascular
Procedure: Endovascular Revascularization — Other would undergo multiple tibialis vessels Endovascular Revascularization

SUMMARY:
This study aims to Compare the outcomes of angioplasty for single tibial vessel occlusion versus multiple tibial vessel occlusions in patients with critical limb ischemia. Assess the effectiveness and safety of angioplasty in treating different extents of tibial vessel occlusions. Evaluate the impact of angioplasty on limb salvage rates, healing of ischemic wounds, and overall clinical improvement in patients with CLI.

DETAILED DESCRIPTION:
This study demonstrates that in patients with chronic limb-threatening ischemia (CLTI), revascularization resulting in the patency of multiple tibial vessels is associated with significantly superior clinical outcomes compared to single-vessel patency. While both strategies were equally safe and technically feasible, the multiple-tibial-vessel (MTV) group achieved perfect limb salvage, higher primary patency, lower restenosis rates, and significantly better wound healing at six months. These findings underscore the importance of robust tibial runoff, supporting the "angiogenic reserve" concept where multiple patent vessels provide redundant perfusion pathways that enhance the durability of revascularization and promote tissue repair. Consequently, when anatomically feasible, treatment strategies should prioritize the establishment or preservation of multi-vessel tibial outflow to optimize limb salvage and functional recovery in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Patients with:

Rutherford Class 5 and 6 Single or multiple occlusive infrapopliteal vessel lesions In-flow vessel (superficial femoral artery and popliteal artery) free from flow-limiting lesion or in-flow lesion correction with bypass or endovascular intervention during index procedure.

Exclusion Criteria:

* Patients with:

Prior vascular intervention in target limb Technical/hemodynamic failure inflow occlusive disease. Patient with allergy to the contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-09 (Actual)

PRIMARY OUTCOMES:
Salvageable of limb(( patients don't need for major amputation )) sabe limb from major amputation | 2years
  Salvageable of limb

CONTACTS AND LOCATIONS:
Overall Officials: Ali Mahmoud Galal, MD of vascular surgery, Study Chair — Aswan University
Locations (1):
- Aswan university hospitals, Aswān, Aswan Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code